CLINICAL TRIAL: NCT04447209
Title: Dietary Diversity of Young Children During CoVID-19 Outbreak: A Longitudinal Study
Acronym: CoDDYC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Lucy Lum Chai See, Professor, University of Malaya
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020410-8500
Record Dates: First submitted 2020-06-17; First posted 2020-06-25 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Dietary Diversity
Keywords: Dietary diversity; micro-nutrient adequacy; young children; urban settings; consumption of sugar sweetened foods and beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child Health Clinic (CHC) (No Intervention): Control arm - Receives dietary counseling but not given food basket.
- Community Children (Experimental): 2-weekly food basket consisting of fresh or minimally processed foods in addition to dietary counseling
  Interventions: Other: 2-weekly Food baskets

INTERVENTIONS:
Other: 2-weekly Food baskets — 2 weekly Food basket containing fresh foods or minimally processed foods.
  Arms: Community Children

SUMMARY:
The 2019-2020 coronavirus pandemic has had far-reaching consequences beyond the spread of the disease. Quarantine measures during a public health pandemic can be particularly detrimental to urban poor families and affect the dietary diversity and food security. This can disproportionately affect young children aged 6 and below, and severely impact those <2 years. Sudden unemployment may result in an unexpected reduction in income that will place pressure on daily budgets for food. Children of families may not have access to foods of adequate diversity that will enable them to meet their macro and micronutrient requirements for growth and development, especially during the Movement Control Order (MCO). The study plans to monitor and evaluate dietary diversity in young children's food intake after the MCO and use the collected information to direct targeted food aid to address observed macro- and micronutrient deficiencies among the urban vulnerable group.

DETAILED DESCRIPTION:
Children are the future to our society. The first thousand days of life, starting from conception till one's second birthday is a critical period of cognitive and physical development. It is the most sensitive period where brain development is most receptive to positive nutrition. Any form of malnutrition, especially during this golden time frame, can lead to irreversible effects to growth, health, education and future career attainment to our potential leaders, which in turn can be a barrier to human development.

The CoVID outbreak is a unique period in recent human history where drastic public health measures such as MCO for an extended period of time has to be implemented nation-wide. These measures have untold severe consequences on the food security of the vulnerable urban group, in particular the young children whose brains require diverse micronutrients to support the rapid growth. These micronutrients can only be obtained from a daily diet that is equally diverse, especially from fresh vegetables and fruits which will be short in supplies. These perishable food items are not usually included in food aids, thus the child may have to subsist on staple-rich diet which are energy-dense but nutrient-poor. These dietary practices are associated with negative health outcomes. Thus by monitoring dietary diversity of the children, we hope to better inform food aid organisations to consider the inclusion of healthier food options to prevent micronutrient deficiencies.

ELIGIBILITY:
Inclusion Criteria:

* All well-children aged between 6 months and 6 years

Exclusion Criteria:

* Children with chronic illnesses

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Minimal Dietary Diversity (MDD) of more than 5 food groups in 24 hours | At study completion, an average of 9 months.
  Number of food groups in 24 hours
Consumption of fruits and vegetables, pre and post-intervention | At study completion, an average of 9 months.
  percentage of population consuming fruits and vegetables, pre and post-intervention
Consumption of sugar-sweetened foods and beverages, pre and post-intervention | At study completion, an average of 9 months.
  percentage of population consuming sugar-sweetened foods and beverages, pre and post-intervention
Height and Weight z-scores, pre and post-intervention | At study completion, an average of 9 months.
  Malnutrition

SECONDARY OUTCOMES:
Blood hemoglobin in children at the start of study and 4 months later | At study completion, an average of 9 months.
  Change in gram/L
Serum ferritin in children at the start of study and 4 months later | At study completion, an average of 9 months.
  Change in microgram/L

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Y Jalaludin, MBBS MPaeds, Study Director — University of Malaya Medical Center
Locations (1):
- University of Malaya Medical Center, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
We will share demographic data of subject and family, baseline anthropometric measurements as well as dietary diversity of children in various locales

REFERENCES:
- [Background] World Health Organization. Indicators for assessing infant and young child feeding practices Part 1: Definitions. Geneva: WHO; 2008
- [Background] Working Group on Infant and Young Child Feeding Indicators. Developing and validating simple indicators of dietary quality of infants and young children in developing countries: Additional analysis of 10 data sets. Report submitted to: the Food and Nutrition Technical Assistance (FANTA) Project/Academy for Educational Development (AED), July 2007
- [Background] Kennedy GL, Pedro MR, Seghieri C, Nantel G, Brouwer I. Dietary diversity score is a useful indicator of micronutrient intake in non-breast-feeding Filipino children. J Nutr. 2007 Feb;137(2):472-7. doi: 10.1093/jn/137.2.472. PMID 17237329
- [Background] Cusick SE, Georgieff MK. The Role of Nutrition in Brain Development: The Golden Opportunity of the "First 1000 Days". J Pediatr. 2016 Aug;175:16-21. doi: 10.1016/j.jpeds.2016.05.013. Epub 2016 Jun 3. No abstract available. PMID 27266965
- [Background] Steyn NP, Nel JH, Nantel G, Kennedy G, Labadarios D. Food variety and dietary diversity scores in children: are they good indicators of dietary adequacy? Public Health Nutr. 2006 Aug;9(5):644-50. doi: 10.1079/phn2005912. PMID 16923296
- [Background] World Health Organization, Geneva. 2017; Global Nutritional Monitoring Framework: Operational guidance for tracking progress in meeting targets for 2025